CLINICAL TRIAL: NCT01533493
Title: Memantine for Executive Dysfunction in Adults With ADHD: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: The American Professional Society of ADHD and Related Disorders (APSARD) (Unknown)
Responsible Party: Principal Investigator, Joseph Biederman, MD, Chief, Clinical and Research Programs in Pediatric Psychopharmacology and Adult ADHD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012P000301
Record Dates: First submitted 2012-02-08; First posted 2012-02-15 (Estimated); Results first posted 2014-02-21 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-03

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD); Executive Function Deficits (EFD)
Keywords: ADHD; Executive Function; Namenda; Concerta
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Memantine; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects randomized to receive memantine-matched placebo in addition to open-label OROS-Methylphenidate
  Interventions: Drug: Placebo; Drug: OROS-Methylphenidate
- Memantine (Active Comparator): Subjects randomized to receive memantine in addition to open-label OROS-Methylphenidate
  Interventions: Drug: Memantine Hydrochloride; Drug: OROS-Methylphenidate

INTERVENTIONS:
Drug: Placebo — Memantine-matched placebo will be prescribed following approved FDA dosing guidelines for Alzheimer's dementia, beginning at 5mg in AM and increasing in BID doses by 5mg weekly to a maximum dose of 10mg BID.
  Arms: Placebo
Drug: Memantine Hydrochloride — Memantine will be prescribed following approved FDA dosing guidelines for Alzheimer's dementia, beginning at 5mg in AM and increasing in BID doses by 5mg weekly to a maximum dose of 10mg BID.
  Other Names: Namenda
  Arms: Memantine
Drug: OROS-Methylphenidate — OROS-Methylphenidate will be openly prescribed, starting with an initial dose of 36mg/day and titrated to optimal response to a maximum daily dose of 1.3mg/kg or 108mg/day, whichever is lower, according to clinician judgment. During titration, dose will be increased on a weekly basis in 36mg/day increments. The dose may be reduced by 18 or 36mg/day increments if adverse effects occur or if the subject discontinues treatment.
  Other Names: OROS-MPH; Concerta

SUMMARY:
This is a 12-week clinical trial evaluating the efficacy and safety of memantine hydrochloride (Namenda) in the treatment of executive function deficits (EFDs) in adults with Attention Deficit Hyperactivity Disorder (ADHD) receiving open-label treatment with OROS-Methylphenidate (OROS-MPH, Concerta). The study aims to examine the effects of treatment with memantine on ADHD symptoms. Following screening procedures, memantine is prescribed in randomized, double-blind fashion (equal chance of medication or placebo) for 12 weeks, along with open-label OROS-MPH (everyone receives medication).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults ages 18-50 years
2. A diagnosis of childhood onset ADHD, according to the Diagnostic and Statistical Manual of Mental Disorder, Fourth Edition (DSM-IV) based on clinical assessment
3. A score of 20 or more on the Adult ADHD Investigator Symptom Report Scale (AISRS)
4. EFDs as established by at least 2 abnormal (>65) subscales of BRIEF-A

Exclusion Criteria:

1. A history of non-response or intolerance to methylphenidate at adequate doses as determined by the clinician
2. A history of non-response or intolerance to memantine at adequate doses as determined by the clinician
3. Pregnant or nursing females
4. A history of clinically unstable or significant other psychiatric conditions including suicidality, homicidality, bipolar disorder, psychosis, or current tic disorder, as judged by the clinician
5. History of narrow angle glaucoma
6. Current (within 3 months) DSM-IV criteria for substance abuse or dependence
7. Medical condition or treatment that will either jeopardize subject safety or affect the scientific merit of the study, including cardiovascular disease, hypertension, history of renal or hepatic impairment, organic brain disorders, or history of seizure disorder.
8. Abnormal hematological or metabolic parameters
9. IQ < 80
10. Current use of any psychotropic medication
11. Lack of facility with the English language
12. Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 33 participants enrolled, 26 were randomized to receive the treatment. The remaining 7 participants were either lost to follow-up after signing consent (n=3) or withdrew consent before being randomized (n=4)
Groups:
- Memantine: Subjects randomized to receive Memantine in addition to open-label OROS-Methylphenidate
  Memantine Hydrochloride : Memantine will be prescribed following approved FDA dosing guidelines for Alzheimer's dementia, beginning at 5mg in AM and increasing in BID doses by 5mg weekly to a maximum dose of 10mg BID.
  OROS-Methylphenidate : OROS-Methylphenidate will be openly prescribed, starting with an initial dose of 36mg/day and titrated to optimal response to a maximum daily dose of 1.3mg/kg or 108mg/day, whichever is lower, according to clinician judgment. During titration, dose will be increased on a weekly basis in 36mg/day increments. The dose may be reduced by 18 or 36mg/day increments if adverse effects occur or if the subject discontinues treatment.
- Placebo: Subjects randomized to receive memantine-matched placebo in addition to open-label OROS-Methylphenidate
  Placebo : Memantine-matched placebo will be prescribed following approved FDA dosing guidelines for Alzheimer's dementia, beginning at 5mg in AM and increasing in BID doses by 5mg weekly to a maximum dose of 10mg BID.
  OROS-Methylphenidate : OROS-Methylphenidate will be openly prescribed, starting with an initial dose of 36mg/day and titrated to optimal response to a maximum daily dose of 1.3mg/kg or 108mg/day, whichever is lower, according to clinician judgment. During titration, dose will be increased on a weekly basis in 36mg/day increments. The dose may be reduced by 18 or 36mg/day increments if adverse effects occur or if the subject discontinues treatment.
Period: Overall Study
Arm/Group | Memantine | Placebo
Started | 12 | 14
Completed | 7 | 11
Not Completed | 5 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Memantine | Placebo | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 14 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.25 (9.77) | 38.43 (10.57) | 36.5 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 5 | 7 | 12
Region of Enrollment [Number; unit: participants]
  United States | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Global Executive Composite T-Score on the Behavior Rating Inventory of Executive Function-Adult (BRIEF-A)
Description: This is a 75-item checklist with a large normative sample, internal consistency, test-retest reliability, inter-rater reliability, and external and concurrent validity, divided into nine empirically and theoretically derived and T-scored subscales: Inhibit, Shift, Emotional Control, Self-Monitor, Initiate, Working Memory, Plan/Organize, Task Monitor, and Organization of Materials. Example item: "I make careless errors when completing tasks." Items are rated 1 "Never," 2 "Sometimes," or 3 "Often." The Global Executive Composite (GEC) Score is calculated by totaling all items on the scale. GEC T-scores range from 34-108, with higher scores indicating more difficulties with executive function.
Time Frame: baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: percentage change from baseline score
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 12 | 14
percentage change from baseline score | -24 (0.169) | -21 (0.132)

ADVERSE EVENTS:
Time Frame: Adverse events were collected weekly, up to 12 weeks.
Arm/Group | Memantine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 10/12 | 13/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Memantine (N=12) | Placebo (N=14)
Anxiety (Psychiatric disorders) | 2 (4) | 2 (2)
Appetite Decrease (Metabolism and nutrition disorders) | 5 (10) | 8/12 (18)
Chest discomfort (Cardiac disorders) | 0 (0) | 2 (2)
Dizziness (General disorders) | 2 (3) | 0 (0)
Dry Mouth (General disorders) | 6 (19) | 6 (8)
Fatigue (General disorders) | 4 (6) | 3 (10)
Forgetting (Psychiatric disorders) | 1 (1) | 2 (2)
Head discomfort (General disorders) | 1 (2) | 3 (5)
Headache (General disorders) | 6 (9) | 2 (2)
Heart Palpitations (Cardiac disorders) | 4 (9) | 4 (12)
Increased Intoxication (General disorders) | 2 (2) | 0 (0)
Insomnia (General disorders) | 3 (4) | 6 (7)
Irritable (Psychiatric disorders) | 2 (3) | 2 (3)
Jittery (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (7)
Nausea (Gastrointestinal disorders) | 2 (4) | 1 (4)
Perceptual Change (Psychiatric disorders) | 2 (2) | 0 (0)
Sweaty Palms (General disorders) | 2 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No